CLINICAL TRIAL: NCT01166815
Title: A Randomized, Double Blind, Controlled Study to Determine the Efficacy of Zinc Supplementation on Diarrhea Incidence in an Adult Population in Western Kenya.
Brief Title: Zinc Supplementation to Reduce Diarrhea Rates in Adults in Western Kenya.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: LTC Maria Bovill, US Army Medical Research Unit - Kenya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: USARIEM C07-04; WRAIR 1332 (Other: Walter Reed Army Institute of Research); KEMRI 1332 (Other: Kenya Medical Research Institute)
Record Dates: First submitted 2010-07-19; First posted 2010-07-21 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2010-07

CONDITIONS: Diarrhea; Malaria
Keywords: diarrhea morbidity; malaria incidence; zinc supplementation
MeSH Terms: conditions — Diarrhea; Malaria | interventions — Zinc Sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zinc supplemented (Active Comparator): Volunteers will be randomly assigned to either receive zinc sulphate supplements (20 mg/capsule) or a placebo containing no zinc. Maltodextrin serves as the carrier. Bulk boxes will identify the products as "A" and "B".
  Interventions: Dietary Supplement: Zinc sulphate
- Placebo (Placebo Comparator): Volunteers will be randomly assigned to either receive zinc sulphate supplements (20 mg/capsule) or a placebo containing no zinc. Maltodextrin serves as the carrier. Bulk boxes will identify the products as "A" and "B".
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Zinc sulphate — Volunteers will be randomly assigned to either receive zinc sulphate supplements (20 mg/capsule) or a placebo containing no zinc. Maltodextrin serves as the carrier. The manufacturer is Tishcon Corporation, Westbury, NY.
  Arms: Zinc supplemented
Other: Placebo — Volunteers will be randomly assigned to either receive zinc sulphate supplements (20 mg/capsule) or a placebo containing no zinc. Maltodextrin serves as the carrier. The manufacturer is Tishcon Corporation, Westbury, NY.
  Arms: Placebo

SUMMARY:
Zinc deficiency is prevalent in children in developing countries. Zinc-supplementation is proven to reduce the duration and severity of childhood diarrhea in randomized controlled trials. However, despite this evidence, its efficacy to reduce diarrhea morbidity in adults remains unknown. The main objective of this study is to determine the efficacy of Zn-supplementation on diarrhea incidences in a vulnerable adult population. The study will be carried out in Kombewa division, Kisumu District and will involve 500 adults aged 18-55 years. They will be randomly assigned to receive Zn supplement (or placebo) on a daily basis over a 3 month period. Morbidity information will be collected daily for 4 months, while anthropometric measures and laboratory data will be obtained at study onset, end of supplementation and study conclusion. In addition, HIV and malaria tests will be carried out during the study as they are important confounders. The significant differences in diarrhea incidence between the Zn-group and the placebo-group will be determined using SPSS. The results are expected to provide the scientific basis and common pathway for development of an anti-diarrheal supplement for vulnerable populations such as environmental refugees, deprived and displaced persons, and troops prior to deployment.

DETAILED DESCRIPTION:
Diarrhea has been a major cause of morbidity, hospitalization, and loss of duty days for military personnel for centuries. In fact, diarrheal illness is the most common medical problem for U.S. troops during operational deployment. Soldiers are especially prone to diarrhea because of travel, consumption of locally procured foods (including raw vegetables and poorly-cooked meat products) and the use of nonpotable water, or ice. High rates of occurrence continue to be reported in soldiers deployed to recent conflicts. Furthermore, high morbidity rates from enteric disease have been reported by other military forces in areas of current combat operations: up to 53%-69% of Soviet troops had major gastrointestinal infections during the Afghanistan war, and up to 69% of British troops and 36% of Australian troops reported diarrhea in Iraq during Operation Safe Haven in 1991.

The region of sub-Saharan Africa, where the proposed study would be conducted, is uniquely positioned for anti-diarrheal research that can offer answers to problems of the civilian population, displaced persons and deployed soldiers or workers in remote areas. Diarrheal disease is the 4th leading cause of out-patient morbidity in Kenya, accounting for almost 5% of all new outpatient cases, with a higher prevalence in Nyanza Province - 5.4% to 7.1% of total new cases. Kisumu lies in the Nyanza Province in western Kenya, bordering Lake Victoria and populated by the Luo ethnic group. Nyanza is one of Kenya's most impoverished provinces with one of the nation's lowest immunization rates, highest infant mortality and highest prevalence of HIV (35% among adults 15-49 years old in 2000, as compared to 14% nationally). Malnutrition is common; endemic diseases include malaria, leishmaniasis, tuberculosis and schistosomiasis.

Scientists from the Centers for Disease Control and Prevention (CDC) have reported on the species of bacterial pathogens isolated from diarrhea patients in the Kisumu area: the bacterial isolates were similar to those reported in U.S. soldiers (44% Shigella; 30% Campylobacter; 14% Salmonella). However, most of the isolates (51%) were not susceptible to their antimicrobial treatment. The study by Brooks et al. (2003), reported that more than 90% of the isolates (excluding Campylobacter) were resistant to trimethoprim-sulfamethoxazole and tetracycline, and more than 80% were resistant to ampicillin.

If this alarming trend persists, and drug-resistant bacteria are identified in civilian populations, gains in disease control strategies already deployed will not be achieved, and in case of deployed members of the military or workforce, mission-impact may be severely compromised. Thus, we propose that the Kombewa Clinical Research Center (KCRC), located outside of Kisumu, would allow for testing of a novel anti-diarrheal treatment, specifically dietary zinc (Zn), in antibiotic-resistant bacteria with potential benefits to not only the deployed U.S. military and western Kenyan populations, but also other populations in Africa. Populations living in the Kombewa area will serve as potential study volunteers because of the high prevalence of antibiotic-resistant diarrhea in adults in this region.

This study will build upon the proven concept that Zn-supplementation, as an adjunct to oral rehydration, is highly protective against diarrhea in children. The results are expected to provide the scientific basis and common pathway for development of a commercially viable, multivalent, food-based, anti-diarrheal supplement for vulnerable populations such as troops prior to deployment, deprived and displaced persons. Based on a successful outcome, we would expect to attract commercial support for a final micronutrient formulation suitable for field use and expanded efficacy evaluation in pivotal studies for support of licensure. An anti-diarrheal product for adults will fill an important military, refugee population need and have dual use in the civilian sector.

The benefits of maintaining adequate zinc status in populations in tropical areas and more so displaced populations such refugees and deployed soldiers are probably not limited to the disease states discussed here. Roles for Zn have been described for other important issues facing the soldier and populations in the tropics especially children, including cutaneous leishmaniasis, malaria, pneumonia, wound healing, cognitive function and behavior, and night vision. Because of these important roles for Zn in maintaining health and fighting disease, maintaining adequate Zn levels and supplementing with Zn in some cases, should be considered when formulating diets for resource deprived populations, displaced people and the modern deployed soldiers.

The primary objective of the study is to determine the incidence of diarrhea in zinc vs. placebo-supplemented adults; secondary objectives include: determining the time to diarrhea onset in both groups; determining the duration of each diarrhea episode in both groups; and determining the number of loose stools per day per episode of diarrhea in both groups. Tertiary objectives include determining the nutritional status of the study population by use of anthropometric measurements and micronutrient assays; determining the incidence of malaria in zinc vs. placebo-supplemented adults; and determining if HIV infection is a confounding factor in the outcome of diarrhea incidences following zinc supplementation in adults.

Hypotheses

1. There is no statistically significant difference in the incidence of diarrhea in adults when given Zn supplementation as compared to placebo over a three month period. We will determine the incidence of diarrhea in both the Zn and placebo arms of the study. This will be accomplished from self-reported incidence of volunteers collected by health workers at the field stations or at the subject's home.
2. The time to diarrhea onset will not be significantly different in the Zn supplemented study arm as compared to the placebo study arm. We will determine the number of days from the study start (this will be after a two week period of volunteers receiving either Zn supplements or placebo) until onset of diarrhea in both the Zn and placebo arms of the study. This will be accomplished from self-reported data of volunteers collected by health workers at the field stations or at the subject's home.
3. The duration of each diarrhea episode will not be significantly different in the Zn-supplemented study arm as compared to the placebo study arm. We will determine the number of days of each diarrhea episode in both the Zn and placebo arms of the study. This will be accomplished from self-reported data of volunteers collected by health workers at the field stations or at the subject's home.
4. The number of loose stools per day per episode of diarrhea will not be significantly different in the Zn-supplemented study arm as compared to the placebo study arm. We will determine the number of number of loose stools per day per episode of diarrhea in both the Zn and placebo arms of the study. This will be accomplished from self-reported data of volunteers collected by health workers at the field stations or at the subject's home.
5. The incidence of malaria will not be significantly different in Zn vs. placebo-supplemented adults. We will determine the incidence of malaria in both the Zn and placebo arms of the study. This will be accomplished using the results from the malaria blood smears collected during the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 55 years of age
* Written informed consent obtained from the volunteer in Dholuo, Kiswahili or English.
* Available to participate for the study duration (approximately five months)
* Negative pregnancy test at screening and study start
* Not taking any vitamin/mineral supplements for the last 2 months prior to onset of the study.

Exclusion Criteria:

* Profound clinical evidence of current immunosuppression or evidence of active AIDS defining illness
* A family history of congenital or hereditary immunodeficiency
* History of allergic reactions to zinc
* History of any neurologic disorders or seizures
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic, renal functional abnormality, as determined by physical examination or laboratory screening tests
* ALT above normal range: >60 U/L Male; >40 U/L Female
* Creatinine above normal range: >1.5 mg/dL
* Hemoglobin below normal range: <11.0 g/dL Male; <9.5 g/dL Female
* Total White Cell Count below normal range <3.0 x 103/uL Male; <2.5 x 103/uL Female
* Absolute lymphocyte count < 1.0 x 103/uL
* Platelet count below normal range <100 x 103/uL
* Pregnant female (positive pregnancy test) at time of screening or study start
* History of chronic alcohol consumption and/or drug abuse
* Use of any investigational or non-registered drugs or vaccines within 30 days preceding the first dose of the study, or planned use during the study period
* Any chronic drug therapy to be continued during the study period
* Simultaneous participation in any other clinical trial
* Planning to start or unable to discontinue vitamin/mineral supplements other than those supplied by the study
* HIV positive with current Aids defining illness or CD4 count less than 250 cells/mm3
* Any other findings that the investigator feels would increase the risk of having an adverse outcome from participation in the trial
* Persons having diarrhea at the time of enrollment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Actual)
Dates: Start 2007-07; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Determine the incidence of diarrhea in zinc vs. placebo-supplemented adults | Daily, for 104 days
  Diarrhea is defined as 3 or more loose motions within a period of 24 hours. Field workers will visit each subject to record diarrhea morbidity data, daily for 104 days.

SECONDARY OUTCOMES:
Determine the time to diarrhea onset in both groups | Daily, for 104 days
  Daily, field workers will visit each subject to dispense supplement and to record diarrhea morbidity data. The time between day 0 and the first bout of diarrhea will be noted.
Determine the duration of each diarrhea episode in both groups | Daily, for 104 days
  Daily, field workers will visit each subject to dispense supplement and to record diarrhea morbidity data. With diarrhea defined as >2 loose motions within a period of 24 hours, the duration (number of days) of the diarrhea will be recorded.
Determine the number of loose stools/day/episode of diarrhea in both groups | Daily, for 104 days
  Daily, field workers will visit each subject to record diarrhea morbidity data. With each bout of diarrhea, we will record the nuber of loose stools/day.

CONTACTS AND LOCATIONS:
Overall Officials: Maria E Bovill, Dr.PH, Principal Investigator — U.S. Army Medical Research Unit - Kenya (USAMRU-K), Kisumu, Kenya; Mark E Polhemus, MD, Principal Investigator — U.S. Army Medical Research Unit - Kenya (USAMRU-K), Kisumu, Kenya; Lucas Otieno, MB.ChB, Principal Investigator — Kenya Medical Research Institute (KEMRI)/Walter Reed Project (WRP), Kisumu, Kenya; Stella K Apollo, BSN, Study Director — Walter Reed Project (WRP), Kisumu, Kenya
Locations (3):
- United States (2):
  - U.S. Army Research Institute of Environmental Medicine (USARIEM), Natick, Massachusetts
  - U.S. Department of Agriculture, Agricultural Research Service, Grand Forks Human Nutrition Center, Grand Forks, North Dakota
- Kombewa Clinical Research Center, Kombewa, Kisumu West, Kenya

REFERENCES:
- [Background] Scrimgeour AG, Lukaski HC. Zinc and diarrheal disease: current status and future perspectives. Curr Opin Clin Nutr Metab Care. 2008 Nov;11(6):711-7. doi: 10.1097/MCO.0b013e3283109092. PMID 18827574
- [Background] Scrimgeour AG, Condlin ML. Zinc and micronutrient combinations to combat gastrointestinal inflammation. Curr Opin Clin Nutr Metab Care. 2009 Nov;12(6):653-60. doi: 10.1097/MCO.0b013e3283308dd6. PMID 19684516
- [Result] AG Scrimgeour, HC Lukaski, ME Polhemus, L Otieno, SM McGraw, AJ Young, ME Bovill. Effect of Zinc Supplementation on Diarrhea and Malaria Morbidity in Adults in Rural Kenya. FASEB J. 2010 24:538.12
- [Result] AG Scrimgeour, HC Lukaski, ME Polhemus, L Otieno, AJ Young, ME Bovill. Zinc supplementation does not alter plasma trace elements in Kenyan adults FASEB J. 2009 23:922.2.